CLINICAL TRIAL: NCT04007185
Title: Assessing Impact of Surgically-induced Deficits on Patient Functioning and Quality of Life (SIND Study)
Brief Title: Surgically Induced Neurological Deficits in Glioblastomas (SIND Study)
Acronym: SIND
Status: Active, not recruiting | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Stephen J Price, NIHR Career Development Fellow and Hon. Consultant Neurosurgeon, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: SIND-2018; CDF-2018-11-ST2-003 (Other Grant/Funding Number: National Institute of Health Research (NIHR))
Record Dates: First submitted 2019-02-19; First posted 2019-07-05 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Glioblastoma
Keywords: quality of life; cognitive function; visual function; surgery
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour samples will be retained as part of routine care in our Tumour Bank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: 30 patients undergoing biopsy for brain tumour. They have the effect of the tumour but not the impact of surgery. Changes in QoL will inform the RCI measures planned
- Surgery Group: The main test group. This group have been determined by their treating surgeon to undergo a resection of the tumour so will be different from the control arm by undergoing a safe, maximal resection of their tumour
  Interventions: Procedure: Maximal, safe resection of brain tumour

INTERVENTIONS:
Procedure: Maximal, safe resection of brain tumour — Standard surgical resection as part of routine care
  Groups: Surgery Group

SUMMARY:
This study provides a work package for a larger programme of research developing Precision Surgery for Glioblastomas by developing individualised treatment volumes for surgery and radiotherapy. This study will recruit a cohort of patients with tumours in different brain regions and involve imaging pre- and post-operatively to outline the area of 'injury' to normal brain. The investigators will then correlate anatomical disruption with changes in measures of quality of life, visual functioning and visual fields and neuropsychology.

DETAILED DESCRIPTION:
This study aims to explore the effect of surgically induced visual and neuro-cognitive defects on patient functioning and quality of life. The aims of this study are:

1. Understand the impact of surgically induced lesions of visual and limbic pathways on quality of life;
2. Determine anatomical regions and brain networks that lead to deterioration in quality of life;
3. Determine extent of early recovery from surgically-induced lesions.

Patient Assessment: Patients will be assessed using the following tools.

1. Ophthalmological assessment - will include:

   1. Acuity (LogMAR - Logarithm of the Minimum Angle of Resolution);
   2. Colour vision (Ishihara);
   3. Basic eye exam to exclude pre-existing ocular pathology (e.g. papilloedema causing a constricted field/enlarged blind spot);
   4. Monocular (Humphrey) and binocular (Esterman) visual field tests.
2. MR imaging - imaging protocol will include:

   1. Standard, anatomical magnetic resonance imaging (MRI)
   2. Diffusion tensor MRI (DTI) - to allow tractography of white matter pathways and to identify post-operative disruption;
   3. Resting state fMRI (rs-fMRI) - to explore plasticity and effect of surgery on functional networks;
   4. 3d contrast enhanced T1-weighted sequence (for surgical planning).
3. Assessment of visual functioning - using the National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) - this 25 item questionnaire assesses difficulty with activities that require vision and their impact on quality of life.
4. Health related quality of life - will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire -30 (EORTC-QLQ30) with the Brain Tumour 20 module (BN20).
5. Cognitive function - neuropsychological will be performed using the OCS-Bridge cognitive screening battery (https://ocs-bridge.com/about.html) on a tablet computer. It takes up to 30minutes to complete:

   1. The Oxford Cognitive Screen (OCS): assesses language, semantics, orientation, reading, movement, number knowledge, mental flexibility, spatial attention and memory.
   2. Cambridge Attention, Memory and Perception Tests: covers visual acuity, verbal and spatial memory, prospective memory, recognition memory, recognition of emotion and sustained attention.
   3. Patient Health Questionnaire (PHQ-9) and Generalised Anxiety Disorder Assessment (GAD-7): measure anxiety and disturbances of mood.
   4. Cognitive reserve - will be estimated pre-operatively (only) using the Cognitive Reserve Questionnaire (CRq) questionnaire that estimates high, medium and low cognitive reserve.

Timings of assessments will be:

1. Baseline assessment: performed pre-operatively.
2. Early assessment: performed in the immediate post-operative period prior to discharge (within 72 hours of surgery). Imaging performed at this time point will be used to determine anatomical disruption following surgery as described in previous studies.
3. Delayed assessment: before radiotherapy starts (within 6 weeks after surgery) to assess recovery. Time points later than this will be confounded by radiotherapy.

Analysis of Clinical Data:

Visual deterioration will be defined as either deterioration in visual acuity (reduction in LogMAR >0.2), or an increase in visual field loss. Deterioration in the NEI-VFQ25 will be determined by published minimal important clinical differences.

Cognitive deterioration: significant abnormalities in cognition are defined as >2 standard deviations from established data from normal patients.

Changes in quality of life: as the investigators expect undergoing surgery alone may be associated with deterioration in quality of life, using published, minimally important clinical differences may not be valid. Instead the investigators will use the reliable change index (RCI) - this this is an individual's score computed as the difference in the baseline and delayed assessment tests divided by the standard error of the difference of the test calculated from a cohort of patients who have undergone an image-guided biopsy (i.e. underwent surgery under anaesthesia with minimal brain disruption) as control subjects.

MR Image Analysis:

1. Voxel-based lesion-symptom mapping will be used to identify the relationships between the surgical site location assessed on MRI and DTI with deterioration in quality of life using methods described in other studies mapping lesions to language and visual deficits.
2. DTI imaging data will study white matter disruption and will be processed in a number of ways -

   1. Measure metrics of the white matter regions to assess effect of tumour invasion using our previously developed methods,
   2. Tractography of the visual pathways will show injury of these pathways using previously developed repeatable and reproducible methods developed.
3. Resting state functional MRI will assess changes to the integrity of brain functional networks and connections. Analysis will include -

   1. independent component analysis (ICA) to identify resting-state networks;
   2. connectome analysis using graph theory measures that correlate to network efficiency, and
   3. fractal analysis looks at the complexity of blood oxygen level (BOLD) time series as a proxy for the capacity for neuronal processing as a global measure of network disruption.

Objectives and key deliverables: The primary objective will be to assess impact of developing a new, permanent surgically-induced visual or cognitive lesion has on quality of life. This will be achieved by understanding the effect of surgically induced visual/cognitive defects on quality of life. This will be achieved by comparing quality of life and NEI-VFQ25 scores for patients with and without newly developed surgically induced deficits.

Secondary objectives will include:

1. Explore which anatomical/functional regions will lead to deterioration in quality of life, neurocognitive function and NIE-VFQ25 scores. This will be achieved by:

   1. Voxel-based lesion-symptom mapping;
   2. White matter tracts disrupted (from DTI data).
2. Investigate recovery of surgically-induced visual/cognitive deficits. This will be studied by comparing visual and cognitive function between initial post-operative assessment and before starting radiotherapy.
3. Quantifying white matter tract disruption by correlating DTI metrics with development of new visual deficits.
4. Assess impact of cognitive reserve on surgically induced cognitive deficits by assessing cognitive decline with different degrees of cognitive reserve.

The investigators will use the data to explore the impact on surgery and changes in cognition and quality of life with disruption of functional brain networks as an exploratory outcome.

Patient Numbers: By recruiting 21 patients with visual deficits and comparing their mean RCI values with 21 patients without such deficits (as controls), an effect size of 0.8 (large) can be detected with 80% probability in a one-sided test (5% type I error rate). An effect size of 0.6 would be detected with a 60% probability under the same conditions with that sample size. From our pilot study data the investigators assume a 25% rate of visual deficit, and therefore 84 patients need to be recruited as a minimum to achieve the required sample size per group. A further 21 patients with frontal lobe lesions will be recruited to look for cognitive decline, and then (generously) assume a 15% drop out figure, so that the total patient numbers will be 120 for this work-package.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate
* Assessed by a neuroscience multi disciplinary team meeting (MDT) to have a high grade glioma on imaging;
* World Health Organisation Performance Scale (WHO PS 0 or 1);
* Patient suitable for tumour resection where the treating neurosurgeon feels that >90% of the enhancing tumour will be resected.

Exclusion Criteria:

* Pre-existing complete homonymous hemianopia or unilateral blindness or visual problems leading to patient being certified sight impaired (visual acuity of 3/60 to 6/60 with a full field of vision or visual acuity of up to 6/24 with a moderate reduction of field of vision or with a central part of vision that is cloudy or blurry).
* Pre-existing severe psychiatric disease
* Patients who are unsuitable for a contrast-enhanced MRI will be excluded.

Such clinical problems include, but are not limited to:

* MR unsafe metallic implants;
* Claustrophobia;
* Allergy to gadolinium contrast agent;
* History of severe renal impairment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Glioblastoma patients presenting to a single neurosciences MDT
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of new deficit on quality of life | 5 +/- 1 weeks post surgery (delayed assessment as defined above)
  Comparison of quality of life measures (using EORTC QLQ30 with BN20 module scores) for patients with and without newly developed surgically induced deficits. These are standard tools for assessing patient reported quality of life

SECONDARY OUTCOMES:
Anatomical disruption | Within 72 hours of surgery (early assessment as defined above)
  Anatomical disruption will be achieved by:
  1. Voxel-based lesion-symptom mapping;
  2. White matter tracts disrupted (from DTI data).
Recovery of visual deficits | 5 +/- 1 weeks post surgery (delayed assessment as defined above)
  Investigate recovery of surgically-induced visual deficits by comparing visual function between early assessment and delayed assessment (before starting radiotherapy). Definitions of visual deficits have been clearly defined in the protocol. To confirm they are - Visual deterioration will be defined as either deterioration in visual acuity (reduction in LogMAR >0.2), or an increase in visual field loss. Deterioration in the NEI-VFQ25 will be determined by published minimal important clinical differences.
Recovery of cognitive deficits using OCS-Bridge tool | Within 72 hours of surgery (early assessment as defined above)
  Investigate recovery of surgically-induced cognitive deficits (measured using the OCS-Bridge tool) by comparing cognitive function between early assessment and delayed assessment. Definitions of cognitive deficits are defined as >2 standard deviations from established data from normal patients.
Quantifying white matter tract disruption | 5 +/- 1 weeks post surgery (delayed assessment as defined above)
  Quantifying white matter tract disruption by correlating DTI metrics with development of new visual deficits. This will be made by comparing visual field deficits (defined as the angle of field loss at delayed assessment compared to baseline) with extent of white matter disruption on DTI (defined from changes in DTI from baseline to early assessment).
Impact of deficits on overall survival | Developing a deficit/not developing deficit will be classified at 6 weeks of surgery (pre-RT). Overall survival figures will be followed until the death of the patient or six months from the last patient undergoing their post-RT assessment.
  Explore impact of new visual and cognitive deficit has on overall survival (defined as date of death from any cause, measured in weeks, assessed up to 3 years post-operatively), compared to patients that don't develop these deficits

OTHER OUTCOMES:
Cognitive reserve | 5 +/- 1 weeks post surgery (delayed assessment as defined above)
  Patients will be divided at baseline into three categories of cognitive reserve using the CRq questionnaire that estimates high, medium and low cognitive reserve. We will correlate these categories with changes in cognitive assessments using the OCS-Bridge tool.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Price, PhD FRCS, Principal Investigator — University of Cambridge
Locations (1):
- Stephen Price, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This is being explored as part of a United Kingdom's Cancer Research UK initiative